CLINICAL TRIAL: NCT07112352
Title: Healthy Ageing: a Feasibility Study to Evaluate Digitally-enabled Ways to Support Healthy Ageing
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 7596188
Record Dates: First submitted 2025-07-09; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Frailty; Older Adults (65 Years and Older); Digital Health Intervention; Feasibility Studies
Keywords: digital health intervention; frailty; older adults (65 years and older); Feasibility study; healthy habit
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Other): Standard care using National Health Service (NHS) guidance on Healthy Ageing for older adults for 6 months.
  Interventions: Other: Control
- Smart devices with Personalised data feedback and habit coaching (Experimental): Participants use smart devices (smartwatch and sleep mat) with a bespoke 'Healthy Habits' application with three healthy habit coaching and data feedback modules focused on active minutes, steps and sedentary time, viewable on a tablet for 3 months. The 'Healthy Habits' application is uninstalled after 3 months and participants will be taught how to use standard 'Withings' application to view their data.
  Interventions: Combination Product: Smart devices with Personalised data feedback and habit coaching
- Smart devices with data feedback (Active Comparator): Smart devices (smartwatch and sleep mat) with a standard off-the-shelf data feedback application ("WithingsTM App") providing generalised data feedback from the participant's smartwatch and sleep mat, viewable on a tablet for 6 months.
  Interventions: Device: Smart devices with data feedback

INTERVENTIONS:
Combination Product: Smart devices with Personalised data feedback and habit coaching — Smart devices (smartwatch and sleep mat) with a bespoke 'Healthy Habits' application with three healthy habit coaching and data feedback modules, focused on active minutes, steps and sedentary time, viewable on a tablet.
  Arms: Smart devices with Personalised data feedback and habit coaching
Device: Smart devices with data feedback — Smart devices (smartwatch and sleep mat) with a standard off-the-shelf data feedback application ("WithingsTM App") providing generalised data feedback from the participant's smartwatch and sleep mat, viewable on a tablet for 6 months.
  Arms: Smart devices with data feedback
Other: Control — Standard care where they will be signposted to National Health Service (NHS) guidance on Healthy Ageing for older adults.
  Arms: Control

SUMMARY:
The goal of this clinical trial is to learn if it is feasibility to conduct a trial of two digitally-enabled interventions that support older adults to adopt healthy behaviours. It will also learn about the safety of this digital intervention. The main questions it aims to answer are

* How acceptable and feasible are the trial, intervention and control groups in assessing outcomes
* What is the estimated effect of the interventions? Researchers will compare Smart devices with a bespoke 'Healthy Habits' application and three healthy habit coaching and data feedback modules, to a group with smart devices and standard off-the-shelf feedback application, to a control group that will receive an education leaflet to adopt healthy behaviours.

Participants will:

* Use sensors and the 'Healthy Habits' application for 3 months followed by standard application for 3 months, or sensors and standard application for 6 months, or control
* Either home visit or in-centre visit once every 3 months for assessments and online health questionnaires
* Complete daily diary of any healthcare use

DETAILED DESCRIPTION:
Frailty is defined as a clinical state manifesting in a reduced capacity to tolerate physiological stressors. This is associated with increased usage of healthcare, healthcare costs and reduced quality of life. This study aims to assess the feasibility of conducting a definitive trial comparing two digitally-enabled interventions that support older adults to adopt healthy behaviours compared to a control. Feasibility will be broken down into trial, intervention and control feasibility. The secondary objectives are preliminary estimation of effect size from the interventions and observation of any persistence effect.

This is a three-arm parallel group non-blinded randomised feasibility trial which involves community-dwelling older adults who are 65 years old and above who are pre-frail as defined by Fried Frailty. Participants are recruited from the community setting.

Potential participants are invited to complete an eligibility questionnaire and screened for eligibility. If eligible, they are consented to participate in the study for six months. On receipt of their consent form, they are randomised into three groups. The groups are A: smart devices with personalised data feedback and habit coaching, B: smart devices with data feedback and a Control group with standard care. Group A will use Smart devices (smartwatch and sleep mat) with a bespoke 'Healthy Habits' application and four healthy habit coaching and data feedback modules focused on active minutes, steps and sedentary time, viewable on a tablet. These modules were co-designed and chosen with participants during a previous Design and Feasibility study. At the end of three months, the application is uninstalled and participants continue to use their smart devices with data feedback.

Participants randomised to Group B will use smart devices (smartwatch and sleep mat) with standard off-the-shelf data feedback application ("WithingsTM App") providing generalised data feedback from the participant's smartwatch and sleep mat, viewable on a tablet for 6 months. Participants randomised to the control group will receive standard care where they will be signposted to the NHS guidance on Healthy Ageing for older adults for six months. Participants will undertake baseline, three and six months online and in-person health assessments and blood test. Participants in Groups A and B will be for feedback about their experience of the programme.

ELIGIBILITY:
Inclusion Criteria:

* • Older adults (age ≥65)

  * Community-dwelling Adults living at home
  * Living within the London boroughs
  * Willing to engage in an exercise programme
  * On at least one medication
  * Pre-frail on Edmonton-AC and/or FRAIL and PRISMA < 3
  * Clinically assessed to have Fried 1-3 (this is completed at baseline assessment)
  * Has the capacity to provide informed consent
  * Able to speak and understand written English

Exclusion Criteria:

* • Adults less than 65 years old

  * Living outside the London boroughs
  * Living in a nursing home or hospitalised or hospice
  * Not taking any medication (indicating robust frailty status)
  * Significant cognitive impairment due to concerns that cognitive impairment and its causes presents different barriers to engagement and participation with sensors and intervention
  * Individuals with severe limitations in activities of daily living which would prevent active participation in the assessments, interfere with participation in the physical exercise programme
  * Being unable to safely engage in the exercise component for other health-related reasons such as Musculoskeletal or neurological disorders that impair gait speed and balance as these are key outcome metrics
  * Progressive or severe medical illness e.g. acute myocardial infarction in the last 3 months, unstable angina, severe aortic stenosis, uncontrolled orthostatic hypotension, recent bone fracture in the last 3 months, having a life expectancy of less than 24 months, requiring palliative care within the following two years, three or more hospitalisations in the last year
  * Moderate - Severe Depression, Psychiatric disorders which may interfere with their participation in the study
  * Being treated for active cancer
  * Unstable medical conditions or where clinical optimisation required e.g. uncontrolled diabetes.
  * Participating in other clinical studies
  * Unable to participate for 6 months in the study (with 28 days allowed to be away from home)
  * Unable to speak or understand written English

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-07-28 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Adherence (%) | 6 months
  This is assessed as a percentage by comparing the number of days the intervention platform is used versus the total number of days enrolled on the study. This will be assessed among participants in Arms A and B.
Triage effectiveness (%) | 6 months
  Triage effectiveness will be evaluated as a percentage by comparing the number of participants that are pre-frail at at first clinical assessment on Fried Frailty assessment versus total participant population. Fried Frialty is assessed using 5 frailty characteristics and is measured on a scale of 0 (best possible score) to 5 (worst possible score). Pre-frail is defined as a score of 1 or 2.

SECONDARY OUTCOMES:
Recruitment rate (%) | 6 months
  Recruitment rate will be assessed by comparing the number of people enrolled and consented to the study compared to number of people invited stratified by each recruitment channel used.
Recruitment diversity (%) | 6 months
  This is assessed by comparing the number of participants from different demographic groups stratified by ethnicity and gender as compared to participant population.
Changes in inflammatory blood markers (C-creative protein) | 6 months
  Blood samples will be collected to evaluate changes in inflammatory marker in the form of C-Reactive Protein (in mg/mL). The levels at baseline will be compared to samples at 3-month and 6-month assessments.
Changes in inflammatory markers (Interleukin-1 level) | 6 months
  Blood samples are collected to evaluate changes in interleukins-1 (in pg/mL). The levels at baseline will be compared to blood samples taken at three and six-month assesssments.
Changes in inflammatory blood level (cortisol levels) | 6 months
  Blood samples will also be collected to evaluate changes in inflammatory markers. This is measured using cortisol (in pg/mL) where baseline levels will be compared to blood samples taken at three and six months assessments.
Completeness of online triage surveys (%) | 6 months
  Online surveys are sent to participants at triage, baseline, three and six months of the study. Completeness of online triage surveys (in percentage) is assessed by comparing the number of completed triage surveys versus total triage surveys started by participants to understand the acceptability of triage procedure.
Safety of intervention and control groups | 6 months
  This is monitored using a Hazard Log of adverse and serious adverse incidents throughout the study. This outcome is assessed by evaluating the number of adverse and serious adverse events in all 3 groups.
Acceptability of control group | 6 months
  This is measured through qualitative feedback on acceptability of the assessments, information and support provided to participants in the control group collected through verbal and free-text responses at three and six-month visits. These responses will be thematically analysed.
Acceptability of intervention using System Usability Scale - SUS | 6 months
  The acceptability of interventions Arms A and B will be assessed using System Usability Score (SUS). The SUS is a ten-item attitude Likert scale giving a global view of subjective assessments of usability. Scores range from 0 (the worst possible score) to 100 (the best possible score). This is evaluated at three and six months of the intervention.
Acceptability of intervention using Unified Theory of Acceptance and Use of Technology | 6 months
  The acceptability of interventions Arms A and B will be assessed using modified Unified Theory of Acceptance and Use of Technology (UTAUT). Modified UTAUT has 25 components each measured on likert scale of 1 being strongly disagree and 5 being strongly agree. This is a range of 25 (worst possible score) to 125 (best possible score). This is assessed at three and six month feedback surveys
Changes in weight (in kg) | 6 months
  Using Withings Smartscale, weight (in kilograms) at three and six months will be compared to baseline assessment.
Changes in Fried Frailty Score | 6 months
  This will be assessed by comparing Fried Frailty Score at 3 and 6 month assessments compared to score at baseline assessment. Fried Frialty is assesses the presence of five frailty characteristics and is measured on a scale of 0 (best possible score) to 5 (worst possible score).
Changes in sleep (Total Sleep Duration) | 6 months
  This is assessed using Withings Sleepmat for changes in total sleep duration (in hours per day) among participants in Arm A and B. The total sleep duration at 6 months will be compared to baseline period of first 7 days of the study.
Change in sedantary time (in minutes) | 6 months
  Changes in sedentary time (in minutes per day) is measured through a smartwatch. This is assessed by comparing the average daily sedentary time at 3 and 6-months as compared to baseline assessment.
Changes in activity levels (number of active minutes) | 6 months
  This will be assessed by comparing average daily active minutes at 3 and 6 months versy average daily active minutes in baseline period. This is measured in active minutes per day as measured by Withings Smartwatch.
Change in Short physical performance battery | 6 months
  This will be assessed by comparing three and six-month scores of Short Physical Performance Battery versus their baseline assessment score. This is measured using three physical tests in units on a scale of 0 (lowest worst score) to 12 (highest best score).
Change in Gait speed (%) | 6 months
  This will be assessed by comparing percentage change in three and six-month assessment of Gait speed (in metres per second) as compared to baseline assessment. Normal walking speed is measured by measuring the time (in seconds) participants take to complete a distance of 15 feet (4.57metres).
Change in Grip strength (in kg) | 6 months
  This will be assessed by comparing three and six-month assessment of grip strength compared to baseline assessment. This is measured using a hand-held dynamometer of participant's dominant hand. This is measured in kilograms.
Changes in cognition using Mini-Addenbrooke cognitive examination | 6 months
  This will be assessed by comparing the three and six-month assessments of participants' total score on the Mini-Addenbrooke Cognitive Examination compared to their baseline assessment. This is a 5-item questionnaire measured in units on a scale of 0 being the lowest score and 30 being the highest score. Scores of less than or equal 25 indicates cognitive impairment.
Changes in Warwick-Edinburgh mental wellbeing scale | 6 months
  This will be assessed by comparing three and six-month asssessment of participants' Warwick-Edinburgh Mental Wellbeing Scale as compared to their baseline assessment. This is a 14-item questionnaire and is measured units on a scale of 7 (worst possible score) to 35 (best possible score).
Changes in Geriatric depression scale | 6 months
  This will be assessed by comparing three and six-month assessment of Geriatric Depression Scale (short form) with the baseline assessment. This is a 15-item questionnaire measured in units on a scale of 0 (best possible score) to 15 (worst possible score).
Changes in Geriatric anxiety scale | 6 months
  This will be assessed by comparing three and six-month assessment of Geriatric Anxiety Scale (GAS-10) as comparing to their baseline assessment. This is a 10-item questionnaire measured on a scale of 0 (best possible score) to 10 (worst possible score).
Changes in Health-related Quality of Life (Short-form 36) | 6 months
  This will be assessed by comparing three and six-month assessment of Health-Related Quality of Life using Short-form 36 (SF-36) as compared to their baseline assessment. SF-36 is a 36-item questionnaire measured on a scale of 0 (worst possible score) to 100(best possible score).
Changes in patient-generated index of independence | 6 months
  This will be assessed by comparing three and six-month assessment of patient-generated index of independence with their baseline assessment. This is a 3-stage questionnaire where participants self-identify and rank most important activities of daily living which is measured on a scale of 0 (worst possible score) to 10 (best possible score).
Changes in social engagement using Lubben Social Network Scale | 6 months
  Social engagement of participants is assessed using Lubben Social Network Scale (LSNS- 6). This will be assessed by comparing the total score of participants' three and six-month assessment of Lubben's social network scale with their baseline assessment. This is a 6-item questionnaire measured on a scale of 0 (worst possible score) to 30 (best possible score).
Changes in sleep using Geriatric Sleep Questionnaire | 6 months
  Self-reported changes in sleep will be assessed by comparing total score on three and six-month assessment online Geriatric Sleep Questionnaire with their baseline assessment. This is a six-item questionnaire measured on a scale of 6 (best possible score) to 30 (worst possible score).
Changes in Step Count (number of steps per day) | 6 months
  Using the Withings SmartWatch, the average daily steps at 3 and 6 months will be compared with average daily steps during baseline period of the first 7 days.
Engagement with online diaries (%) | 6 months
  This is assessed by comparing the number of daily diary entriees completed online compared with the total daily diary entries completed online for participants in Group A.
Healthcare resource utilisation | 6 months
  This is assessed by number of self-reported episodes of visits to primary, secondary and tertiary healthcare facilities in all three groups during the study. This is assessed in Arm A in their daily diary entries. This is assessed in their 3 and 6-month assessments.
Clinical Record Form (CRF) completeness (%) | 12 months
  This is assessed as a percentage by comparing the number of clinical record forms completed at 3 months, 6 months, 9 months and 12 months compared with the total number of forms requested. These forms are completed by the research team for all participants.
Change in body composition (%) | 6 months
  This is assessed using Withings Smartscale which measures fat mass (in percentage). The Fat mass percentage at baseline assessment will be compared to three and six-month measurements.
Changes in sleep - total snoring duration per night | 6 months
  This is assessed using Withings Sleep mat which records the total duration of snoring. This is assessed by comparing changes as a percentage of the total snoring duration per night during the baseline period of first 7-days compared with total snoring duration per night at 3 and 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Leila Shepherd, MEng, PhD, Principal Investigator — Imperial College London
Locations (1):
- Helix Centre, Institute of Global Health Innovation, Department of Surgery and Cancer, Imperial College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Participants are not consented for data sharing outside team.